CLINICAL TRIAL: NCT03025906
Title: Phenobarbital Versus Valproate for Generalized Convulsive Status Epilepticus in Adults: A Prospective Randomized Controlled Trial in China
Brief Title: Phenobarbital Versus Valproate for Generalized Convulsive Status Epilepticus
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Principal Investigator, Yingying Su, neurology department, Xuanwu Hospital, Beijing
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WEIBANYIZHENGHAN[2012]649
Record Dates: First submitted 2016-11-15; First posted 2017-01-20 (Estimated); Last update posted 2019-07-09 (Actual); Status verified 2019-07

CONDITIONS: Generalized Convulsive Status Epilepticus
MeSH Terms: conditions — Status Epilepticus | interventions — Phenobarbital; Valproic Acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phenobarbital (Experimental): In the PB group, a loading dose of 20 mg/kg (may give an additional 10 mg/kg) begins at a rate of 50 mg/min followed by IV 100 mg q6 h.
  Interventions: Drug: Phenobarbital
- Valproate (Experimental): In the VPA group, a loading dose of 30 mg/kg (may give an additional 15 mg/kg) begins at a rate of 3 mg/kg per min followed by a continuous infusion at a rate of 1-2 mg/kg per hour.
  Interventions: Drug: Valproate

INTERVENTIONS:
Drug: Phenobarbital — In the PB group, a loading dose of 20 mg/kg (may give an additional 10 mg/kg) begins at a rate of 50 mg/min followed by IV 100 mg q6 h.
  Other Names: Luminal
  Arms: Phenobarbital
Drug: Valproate — In the VPA group, a loading dose of 30 mg/kg (may give an additional 15 mg/kg) begins at a rate of 3 mg/kg per min followed by a continuous infusion at a rate of 1-2 mg/kg per hour.
  Other Names: Depakine
  Arms: Valproate

SUMMARY:
Although generalized convulsive status epilepticus (GCSE) is a life-threatening emergency, evidence-based data to guide initial drug treatment choices are lacking in the Chinese population. The investigators conduct this prospective randomized controlled trial to evaluate the relative efficacy and safety of intravenous (IV) phenobarbital (PB) and valproate (VPA) in patients with GCSE.

DETAILED DESCRIPTION:
After the failure of first-line diazepam treatment, patients with GCSE are randomized to receive either IV PB (standard doses, low rate) or VPA (standard). Successful treatment is considered when clinical and electroencephalographic seizure activity ceases. Adverse events following treatment and the neurological outcomes at discharge and 3 months later are also evaluated.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive GCSE patients (after the failure of first-line diazepam treatment) who were admitted in the emergency room or neurocritical care unit in Xuanwu Hospital of Capital Medical University.

Exclusion Criteria:

* Unstable vital signs, such as a systolic blood pressure of <90 mm Hg, a pulse of <60 beats per min, or an arterial blood oxygen saturation of <90%,
* Liver dysfunction (alanine transaminase or total bilirubin of more than twice the normal upper limit),
* Neurologic emergency requiring immediate surgical intervention,
* Pregnancy or breast feeding,
* Hypersensitivity to study drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2017-02-16 (Actual); Primary Completion 2019-10 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients with effective seizure control | One hour after the end of the PB or VPA loading dose
  The primary study endpoint is the number of patients with effective seizure control, defined as a cessation of clinical and electroencephalographic seizure activity within 1 h after administration of the phenobarbital or valproate loading dose. Effective control of GCSE is assessed clinically by one certified neurologist and also confirmed with EEG by one certified electroencephalographer.

SECONDARY OUTCOMES:
Mortality of patients | at 30 days and at 3 months
  Neurologic outcome is assessed both at 30 days and at 3 months by one physician unaware of the therapeutic assignment through a phone interview or scheduled follow-up clinic visit. Mortality of each group is recorded at 30 days and at 3 months, respectively.
Number of patients with post-SE symptomatic epilepsy | 3 months
  Post-SE symptomatic epilepsy at 3 months is analyzed. It is defined as the occurrence of at least 2 unprovoked epileptic seizure occurring not earlier than 4 weeks after termination of SE in those without pre-existing epilepsy.
The relapse rates of SE and nonconvulsive status epilepticus (NCSE) / nonconvulsive seizures (NCS) | in the first 24 h
  The investigators also record the relapse rates of SE and nonconvulsive status epilepticus (NCSE) / nonconvulsive seizures (NCS) in each group in the first 24 h.

OTHER OUTCOMES:
Number of Participants With Adverse Events | From the administration of PB or VPA to 1 week
  Adverse events are recorded as follows: systolic blood pressure lower than 90 mmHg, pulse lower than 50 beats/ min, arrhythmia (except supraventricular tachycardia), respiratory depression (arterial oxygen saturation below 90%, partial pressure of oxygen below 60 mmHg, or partial pressure of carbon dioxide above 60 mmHg), drug-induced liver disease (alanine aminotransferase or total bilirubin increase of more than twice the upper limit of the normal range), elevation of blood ammonia (more than twice the upper limit of the normal range), gastric motility insufficiency, bone marrow suppression (leukocytopenia, neutrocytopenia, thrombocytopenia or anemia), coagulation disorders, or drug-related sedation. The time to record adverse events is from the administration of PB or VPA to 1 week.

CONTACTS AND LOCATIONS:
Locations (6):
- China (6):
  - Xuanwu Hospital, Beijing, Beijing Municipality
  - Zhongshan Hospital, Xiamen University, Xiamen, Fujian
  - Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong
  - Xiangya Hospital, Central South University, Changsha, Hunan
  - Xijing Hospital, Shanxi, Xi'an
  - The First People's Hospital of Yunnan Province, Kunming, Yunnan

IPD SHARING:
Plan to Share IPD: Undecided